CLINICAL TRIAL: NCT03144323
Title: The Effectiveness of Electronic Reminders in Improving Intra-oral Elastic Compliance in Orthodontic Patients: A Randomised Clinical Trial
Brief Title: The Effectiveness of Electronic Reminders in Improving Elastic Compliance in Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 209439
Record Dates: First submitted 2017-01-30; First posted 2017-05-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Malocclusion; Compliance, Patient
Keywords: Intraoral elastics
MeSH Terms: conditions — Malocclusion; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group will receive 4 daily electronic reminders via the Calendar app on their mobile phones, reminding them to wear their elastics.
  Interventions: Behavioral: Reminders
- Control group (No Intervention): This group will receive their orthodontic treatment and elastics instructions as normal, without reminders.

INTERVENTIONS:
Behavioral: Reminders — Four reminders will be set on the patient's mobile phone's Calendar-type app, saying "Don't forget to wear your elastics", at 08:00, 13:00, 17:00 and 22:00.
  Arms: Study group

SUMMARY:
Fixed orthodontic appliances in combination with intraoral elastics are a common and effective method use in the orthodontic correction of malocclusions. However, their success is largely dependent on the patient's compliance. Failure to wear the elastics as instructed will reduce efficacy of treatment, ultimately increasing treatment time and potentially producing imperfect alignment of teeth.

The hypothesis tested is that daily electronic reminders via a mobile application can significantly increase patient compliance, thus effectively improving treatment outcomes.

DETAILED DESCRIPTION:
Despite advancements in various aspects of orthodontic treatment, patient compliance remains a critical factor in attaining a successful treatment outcome. More specifically, patient compliance in the use of intraoral elastics is an important component of the treatment plan of certain patients. Failure to wear elastics as directed will ultimately result in increased treatment time, and imperfect alignment of the teeth.

Persuading adolescent orthodontic patients to wear intraoral elastics consistently is difficult in the short appointment times of a typical practice. Studies have shown that adolescents respond at a higher level to a more constant form of communication, as well as a method more closely associated with their generation. As smartphones have become an everyday appliance for most of the general public, mobile applications (apps) have the capability to serve as an effective avenue for communication between doctor and patient. Recent studies in both dentistry and medicine have reported that active reminders via mobile phone improve appointment attendance, adherence to medication schedules, and positive behaviour changes.

The investigators will utilise the "Calendar" app to communicate via daily reminders with patients undergoing orthodontic treatment with fixed appliances and Class II intraoral elastics, and they will measure the improvement in the malocclusion. This will allow study of whether or not electronic reminders can significantly increase compliance.

As more apps are developed, this communication method may have the potential to greatly impact the way orthodontists and patients interact outside of the office. If effective, these apps could become a cornerstone of the compliance efforts of many orthodontic practices. This would benefit both the orthodontist and the patient, as it would decrease time and money spent for both parties as well as reduce the overall sense of frustration felt during extended orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Full fixed appliances with intraoral class II elastics full-time
* Wearing class II elastics for between 6 weeks & 3 months
* Have smartphone with calendar-type app

Exclusion Criteria:

* Orthognathic surgery planned
* Craniofacial disorders

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of elastics used and collected by the participant | 6 weeks, 12 weeks
  Participants from both arms will collect their used elastics in a plastic bag provided, which will be collected at each recall appointment and counted.

SECONDARY OUTCOMES:
Patient's self-reported duration of time spent wearing intraoral elastics | 6 weeks and 12 weeks
  Participants will fill out duration journals between appointments, on which they tick boxes to record how many hours a day they have worn their elastics
Change in participant's jaw relationship, measured on mm scale by difference in overbite, overjet and molar relationship | Baseline, 6 weeks, and 12 weeks
  Clinicians will record these occlusal measurements at each appointment
Clinician-perceived level of compliance of the participant at each appointment, using discrete qualitative scale | Baseline, 6 weeks, and 12 weeks
  Clinicians will record whether they think the patient has been highly, somewhat, or not at all compliant

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bister, Study Director — Guy's and St Thomas's Hospital NHS Foundation Trust; Jadbinder Seehra, Principal Investigator — King's College Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - Guy's Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No